CLINICAL TRIAL: NCT05096364
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Phase II Clinical Study to Evaluate the Efficacy and Safety of AK111 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Phase 2 Study of Efficacy and Safety of AK111 in Subjects With Moderate-to-Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK111-201
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Psoriasis
Keywords: AK111; efficacy; safety
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AK111 Regimen 1 (Experimental): AK111 Regimen 1 - subcutaneous injection every 4 weeks up to 60 weeks
  Interventions: Biological: AK111/Placebo
- AK111 Regimen 2 (Experimental): AK111 Regimen 2 - subcutaneous injection every 4 weeks up to 60 weeks
  Interventions: Biological: AK111/Placebo
- AK111 Regimen 3 (Experimental): AK111 Regimen 3 - subcutaneous injection every 4 weeks up to 60 weeks
  Interventions: Biological: AK111/Placebo
- AK111 Regimen 4 (Experimental): AK111 Regimen 4 - subcutaneous injection every 4 weeks up to 60 weeks
  Interventions: Biological: AK111/Placebo
- Placebo to AK111 (Placebo Comparator): Placebo to AK111-Placebo subcutaneous injection, then 1:1 randomized to AK111 Regimen 3 or Regimen 4 at week 12
  Interventions: Biological: AK111/Placebo

INTERVENTIONS:
Biological: AK111/Placebo — After loading dose, investigational drug was administered subcutaneously up to 60 weeks.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center Phase II clinical study to evaluate the efficacy and safety of AK111 for the treatment of moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center Phase II clinical study to evaluate the efficacy and safety of AK111 in subjects with moderate to severe plaque psoriasis. The study will consist of 4 periods: up to 4 weeks screening period, 12 weeks placebo-controlled period,12 weeks crossover treatment period,44 weeks long-term treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, 18 to 75 years of age
2. Moderate to severe plaque-type psoriasis diagnosed for at least 6 months
3. Moderate-to-severe plaque psoriasis as defined at baseline by meeting all three criteria:

   1. Clinical diagnosis of stable plaque psoriasis with involvement of ≥ 10% body surface area.
   2. Psoriasis area and severity index(PASI) ≥12.
   3. Static Physicians Global Assessment score ≥3.
4. Subjects with a history of an inadequate response, intolerable or medically inappropriate use of systemic therapy and/or phototherapy.
5. Subjects who are women of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 8 months after the last study drug administration.

Key Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type psoriasis.
2. History or evidence of active TB, Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment according to protocol.
3. Positive results of confirmatory serology test for hepatitis B, hepatitis C, HIV or syphilis at screening.
4. History of a serious or systemic infection within 2 months before screening.
5. History of malignancy of any organ system within the past 5 years.
6. Inadequate washout period for prior drug therapy.
7. Previous use of secukinumab, ixekizumab or any other drug that targets IL-17 or IL-17 receptor.
8. Any medical conditions, in the opinion of the Investigator or the Sponsor's medical monitor, would place the subject at risk, interfere with study participation or study results interpretation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve Psoriasis Area and Severity Index (PASI) 90 response or higher at week 12 | At week 12

SECONDARY OUTCOMES:
Proportion of subjects who achieve PASI 75 response or higher at week 12 | At week 12
Proportion of subjects who achieve static Physician Global Assessment (sPGA) 0 or 1 at week 12 | At week 12
Proportion of subjects who achieve PASI 50, PASI 75, PASI 90 and PASI 100 response up to 68 weeks | Baseline to week 68
AK111 concentrations in serum at different time points | Baseline to week 68
Number and proportion of subjects who developed anti-drug antibodies (ADAs) | Baseline to week 68
Change in serum IL-17A level (Pharmacodynamics parameter） | Baseline to week 68
Adverse events (AEs)/serious adverse events (SAEs) | Baseline to week 68

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - AkesoBio Investigative Site 1011, Bengbu, Anhui
  - AkesoBio Investigative Site 1009, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1016, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 1003, Guangzhou, Guangdong
  - AkesoBio Investigative Site 1007, Guangzhou, Guangdong
  - AkesoBio Investigative Site 1012, Chengde, Hebei
  - AkesoBio Investigative Site 1018, Harbin, Heilongjiang
  - AkesoBio Investigative Site 1008, Changsha, Hunan
  - AkesoBio Investigative Site 1013, Yancheng, Jiangsu
  - AkesoBio Investigative Site 1001, Shanghai, Shanghai Municipality
  - AkesoBio Investigative Site 1010, Shanghai, Shanghai Municipality
  - AkesoBio Investigative Site 1002, Hanzhou, Zhejiang
  - AkesoBio Investigative Site 1006, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No